CLINICAL TRIAL: NCT01724151
Title: Effects of Exercise Training in Patients With Mild Cognitive Impairment
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200812152R
Record Dates: First submitted 2010-02-25; First posted 2012-11-09 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy adults: Healthy adults, over 45 years old
- Mild cognitive impairment: subjects with mild cognitive impairment
- Alzheimer's disease: subjects with Alzheimer's disease

SUMMARY:
The proposes of this study are

1. To understand the physical activities of patients with cognitive impairment in Taiwan and construct the validity and reliability of the physical activity questionnaire and actigram in this population.
2. To understand the relation between brain structure (brain tractography and resting state functional MRI) and cognitive and physical functions of patients with cognitive impairment, the capability of activity and social engagement (including quality of life).
3. To understand the efficacy of exercise on the brain structure (brain tractography and resting state functional MRI), cognitive and physical functions, the capability of activity and social engagement (including quality of life) of the patients with cognitive impairment.

The study aims to establish the data base of physical activity of patients with cognitive impairment in Taiwan. We will also analyze the efficacy of exercise with ICF model on physical function, physical activity and social engagements to provide an optimized design of exercise program for patients with cognitive impairment in the future.

DETAILED DESCRIPTION:
There is already evidence that exercise training can delay the progression of dementia. But if the same effect could be seen in patients with cognitive impairment remains unknown. There is an increasing importance of how to delay or prevent the turn over of cognitive impairment patients into dementia in recent years. Thus we propose to investigate the following issues.

1. To understand the physical activities of patients with cognitive impairment in Taiwan and construct the validity and reliability of the physical activity questionnaire and actigram in this population.
2. To understand the relation between brain structure (brain tractography and resting state functional MRI) and cognitive and physical functions of patients with cognitive impairment , the capability of activity and social engagement (including quality of life).
3. To understand the efficacy of exercise on the brain structure (brain tractography and resting state functional MRI), cognitive and physical functions, the capability of activity and social engagement (including quality of life) of patients with cognitive impairment.

The study is a cross sectional study. We recruited 40 cognitive impairment patients from the memory clinic at National Taiwan University Hospital and another 20 healthy controls matched for age and gender. We collected the actigram and physical activity from questionnaire for 7 days and performed the analysis for reliability and validity. We will do correlation analysis with the data with resting state functional MRI and tractography, brain connectivity, and plasma Aβ1-40 and Aβ1-42 amyloid protein.

The study aims to establish the data base of physical activity of patients with cognitive impairment in Taiwan. We will also analyze the efficacy of exercise with ICF model on physical function, physical activity and social engagements to provide an optimized design of exercise program for patients with cognitive impairment in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Above 45 years old and had independent walking ability
2. The MCI is diagnosed basically on Petersen's criteria (Petersen, 2001), CDR score of 0.5 but normal ADL/IADL, and not demented
3. Diagnosis of Alzheimer's disease based on NINCDS-ADRDA criteria for probable AD (McKhann, et al., 1984)

Exclusion Criteria:

* The subjects who had any neurological, musculoskeletal, cardio-pulmonary disorder which would cause gait disorder or cognitive dysfunction such as stroke, Parkinson disease, or arthritis were excluded

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic,community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Walking speed of participants | 1 hour
  Subjects walk through 10m walkway with steady comfortable pace. We record complete duration and calculate walking speed (m/sec)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jang Chiu, Study Chair — Neurology department, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan